CLINICAL TRIAL: NCT03405376
Title: Prospective Trial of Treat and Extend Aflibercept for Macular Edema Secondary to Branch Retinal Vein Occlusion: the PLATON Trial
Brief Title: Prospective Trial of Treat and Extend Aflibercept for Macular Edema Secondary to Branch Retinal Vein Occlusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Min Sagong, Associate Professor, Yeungnam University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YUMC2017-07-056-003
Record Dates: First submitted 2018-01-14; First posted 2018-01-23 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Branch Retinal Vein Occlusion With Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Branch retinal vein occlusion (Experimental): Aflibercept 2mg is injected into the vitreous cavity. Center-involved macular edema secondary to branch retinal vein occlusion for no longer than 3 months (at the screening visit it should be ensured that the subjects will comply with the criterion of ≤ 3 months since onset of macular edema at their scheduled baseline visit)
  Interventions: Drug: Intravitreal aflibercept injection

INTERVENTIONS:
Drug: Intravitreal aflibercept injection — Aflibercept 2mg is injected into the vitreous cavity through the pars plana using 30G needle-attached syringe for branch retinal vein occlusion.
  Other Names: Eylea, VEGF Trap-Eye

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the treat-and-extend regimen extending to 4 months by intervals of 4 weeks using intravitreal aflivercept injection for treatment of macular edema secondary to BRVO.

DETAILED DESCRIPTION:
Retinal vein occlusion (RVO) includes central RVO (CRVO) and branch RVO (BRVO). A highly prevalent retinal vascular disease, RVO is second only to diabetic retinopathy. In CRVO, hemorrhages and edema develop throughout the retina, whereas in BRVO the pathology is more sectoral, involving the portions of the retina drained by the obstructed branch vein. This suggests that increased intraluminal pressure behind the obstruction may lead to transudation of blood cells and plasma into the retina. However, recent studies have demonstrated that although increased venous pressure may be the precipitating event for hemorrhages and edema, increased production of vascular endothelial growth factor (VEGF) occurs early in RVO and is a major contributor to their evolution and persistence. In addition, the high levels of VEGF contribute to progression of retinal nonperfusion and hence retinal ischemia, which may in turn increase production of VEGF, and may explain why some eyes enter a vicious cycle of worsening disease often referred to as conversion to an ischemic RVO.

Treat-and-extend intravitreal anti-VEGF with age related macular degeneration and diabetic macular edema has been reported to offer the opportunity to individual management while minimizing treatment burden and similar visual and anatomical outcomes to those with fixed montly dosing.

Also, small retrospective treat-and-extend intravitreal bevacizumab injection for treatment of BRVO associated macular edema demonstrated similar visual outcomes and number of intravitreal injections as did pro-re-nata treatment with ranibizumab conducted in phase 3 trials but with fewer visits and lower annual medical costs.

The effects of afilbercept have been reported to persist for over 8 weeks in DME and AMD studies. In addition, VIBRANT study also demonstrated that bi-monthly injection of aflibercept showed significant visual improvement in BRVO patients.

In the treat-and-extend studies of RVO, ranibizumab has been extended for up to 4 months at intervals of 2 weeks. But, to our knowledge, there was no prospective study of treat-and-extend regiments with intravitreal aflibercept in treatment naïve patients in BRVO.

ELIGIBILITY:
Inclusion Criteria:

* Center-involved macular edema secondary to BRVO for no longer than 3 months (at the screening visit it should be ensured that the subjects will comply with the criterion of ≤ 3 months since onset of macular edema at their scheduled baseline visit).
* Adult subjects diagnosed with macular edema secondary to BRVO who are scheduled to be treated with intravitreal aflibercept as per investigator's routine treatment practice with the intent to use a T&E regimen after initial treatment.
* Treatment-naïve subjects for macular edema secondary to BRVO.
* Both ischemic and non-ischemic BRVO, which are confirmed by FA at baselin, week 24 and week 72.
* Men and women ≥ 18 years of age.
* Documented BCVA of ETDRS letter score of 73 to 24 letters (Snellen equivalent of 20/40 to 20/320) in the study eye.

Exclusion Criteria:

* Previous PRP or macular laser photocoagulation in the study eye.
* Any prior or concomitant ocular treatment (e.g. anti-VEGF therapy, corticosteroids) in the study eye for macular edema secondary to BRVO, except dietary supplements or vitamins prior to inclusion in the study. Intraocular anti-VEGF treatment is permitted for the treatment of diseases of fellow eye except for those that are specifically excluded.
* Prior systemic anti-VEGF or corticosteroid therapy, investigational or approved, within the last 3 months before the first dose in the study.
* Previous use of intraocular corticosteroids in the study eye at any time or use of periocular corticosteroids in the study eye within 12 months prior to Day 1.
* Any active intraocular, extraocular, and periocular inflammation or infection in either eye within 4 weeks of screening.
* Any history of allergy to povidone iodine.
* Known serious allergy to the fluorescein sodium for injection in angiography.
* Presence of any contraindications indicated in the EU commission/locally approved label for intravitreal aflibercept: hypersensitivity to the active substance intravitreal aflibercept or to any of the excipients; active or suspected ocular or periocular infection; active severe intraocular inflammation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean change of best corrected visual acuity | From baseline to Week 72
  The mean change of best corrected visual acuity from baseline to Week 72 in early treatment diabetic retinopathy letter score

SECONDARY OUTCOMES:
Mean change of best corrected visual acuity | From baseline to Week 24, 52
  The change in mean best corrected visual acuity at baseline as measured by the early treatment diabetic retinopathy letter score
mean change in central macular thickness | From baseline to Weeks 24, 52, and 72
  The mean change in central macular thickness
mean treatment interval between injections | From baseline to Week 72
  The mean treatment interval between injections
gain ≥ 15 letters in best corrected visual acuity | Compared with baseline at Week 24, 52 and 72
  The proportion of subjects who gain ≥ 15 letters in best corrected visual acuity on the early treatment diabetic retinopathy chart
mean treatment interval between injections of ≥ 12 or 16 weeks | From the last actual visit of the initiation phase to Week 72
  The proportion of subjects with a mean treatment interval between injections of ≥ 12 or 16 weeks
who reach 16 weeks treatment interval at any time point | up to 72 weeks
  The proportion of subjects who reach 16 weeks treatment interval at any time point

CONTACTS AND LOCATIONS:
Overall Officials: Min Sagong, MD, Principal Investigator — Yeungnam University Hospital
Locations (5):
- South Korea (5):
  - Min Sagong, Daegu, Deagu
  - Dong-A University Hospital, Busan
  - Maryknoll Medical Center, Busan
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju